CLINICAL TRIAL: NCT03405779
Title: A Pilot Study of a New Ultrasonographic Tool to Assess Regional Pulmonary Strain in Mechanically Ventilated Patients Suffering From Pulmonary Diseases in an Intensive Care Setting.
Brief Title: A New Ultrasonographic Tool to Assess Pulmonary Strain in the ICU
Status: Recruiting | Type: Observational
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Other Study IDs: 17.277
Record Dates: First submitted 2018-01-15; First posted 2018-01-23 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Mechanical Ventilation Complication; Ventilator-Induced Lung Injury
MeSH Terms: conditions — Ventilator-Induced Lung Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: Lung ultrasonography — Mechanically ventilated patients suffering from pulmonary diseases will undergo a lung ultrasonography during their stay in the intensive care unit (ICU)

SUMMARY:
The primary objective of the study is to create a small dataset of regional pulmonary strain values in patients suffering from pulmonary diseases under mechanical ventilation in an intensive care setting.

Hypothesis: The analysis of lung ultrasonographic sequences using speckle-tracking allows the determination of local pleural strain in 4 predetermined pulmonary areas in mechanically ventilated patients suffering from pulmonary diseases.

DETAILED DESCRIPTION:
Mechanical ventilation is frequently used in the intensive care settings. Although essential in many cases, mechanical ventilation can be responsible for ventilator-induced lung injury (VILI). The relationship between mechanical ventilation and VILI has been clearly demonstrated in animals and is highly suspected in humans. The putative mechanism responsible for VILI is excessive pulmonary strain or overdistension. Frequently observed in mechanically ventilated patients, the presence of severe pulmonary disease can increase the risk of overdistension. The development of a tool allowing early detection of pulmonary overdistension would represent a great asset in the prevention of VILI by allowing safer adjustments of mechanical ventilation parameters. Ultrasonographic imaging is a non-radiant, non-invasive technique already available in the intensive care setting. Presently used for cardiac strain measurements, ultrasonography is a promising avenue to assess pulmonary strain.

This pilot study will aim to create a small dataset of local pleural strain values assessed in 4 predetermined pulmonary areas using ultrasonographic imaging in mechanically ventilated patients suffering from pulmonary diseases in the intensive care setting. This dataset will be used to help plan larger scale studies.

Methods:

Intensive care patients under mechanical ventilation will undergo imaging of the pleura at 4 predetermined areas. The sites to be studied will be: the 3rd intercostal space at the mid-clavicular line (left and right side), the 8th intercostal space at the posterior axillary line (left and right side). Three consecutive respiratory cycles at each site will be recorded for subsequent analysis.

Lung ultrasonography will be performed by the principal investigator and a co-investigator using a Terason (Teratech Corporation, Burlington, MA) device and a 12L5 linear ultrasound probe. For each image, the probe will be oriented perpendicularly to the pleura with the pointer towards the participant's head. The beam's focal zone will be positioned at the level of the pleural line.

Using a reference ultrasonographic image, an experienced lung ultrasonographer will segment the pleura. From this image, an algorithm will define a region of interest which will be followed throughout the rest of the images of the video sequence. Thereafter, the algorithm will calculate the various components of pulmonary strain. An experienced technician will visually validate the algorithm's tracking.

ELIGIBILITY:
Inclusion Criteria:

* Adult intensive care patients under mechanical ventilation suffering from a pulmonary disease with a static lung compliance of less than 40 mL/cm H2O.

Exclusion Criteria:

* Obesity (Body Mass Index superior to 30 kg/m2)
* Previous thoracic procedure (chest tube, thoracotomy, thoracoscopy)
* Intra-abdominal pressure inferior to 15 mm Hg (if available)
* Previous participation to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult Intensive care patients under mechanical ventilation suffering from a pulmonary disease.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2018-03-12 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Average absolute lateral deformation | At the end of study on Day 1
  Change in percentage from baseline expiratory value

SECONDARY OUTCOMES:
Cumulated range of absolute lateral deformation | At the end of study on Day 1
  Change in percentage from baseline expiratory value
Average absolute axial deformation | At the end of study on Day 1
  Change in percentage from baseline expiratory value
Cumulated range of absolute axial deformation | At the end of study on Day 1
  Change in percentage from baseline expiratory value
Average von mises | At the end of study on Day 1
  Change in percentage from baseline expiratory value
Average absolute lateral shear | At the end of study on Day 1
  Change in percentage from baseline expiratory value
Cumulated range of absolute lateral shear | At the end of study on Day 1
  Change in percentage from baseline expiratory value

CONTACTS AND LOCATIONS:
Overall Officials: Martin Girard, MD,FRCPC, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre Hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No